CLINICAL TRIAL: NCT03273192
Title: A Randomised, Double-blind, Single-dose, Parallel-group Study in Healthy Subjects to Demonstrate Pharmacokinetic Equivalence of CinnoRA® (Produced by CinnaGen CO.) and Humira® (the Reference Drug, Produced by AbbVie Inc.)
Brief Title: A Study Of CinnoRA (Adalimumab-CinnaGen) And Adalimumab (Humira) In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ADA.CIN.AJ.95 (I-PK)
Record Dates: First submitted 2017-09-03; First posted 2017-09-06 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Bioequivalence; Phase 1
Keywords: healthy subjects; adalimumab; single dose; Phase 1; PK
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CinnaGen adalimumab (Experimental): CinnoRA® (adalimumab auto-injector devices produced by CinnaGen Company) 40 mg/0.8 ml in auto-injector devices A single 40-mg dose of Adalimumab was subcutaneously administered to healthy subjects.
  Interventions: Drug: Adalimumab
- AbbVie adalimumab (Active Comparator): Humira® (adalimumab auto-injector devices produced by AbbVie Company) 40 mg/0.8 ml in auto-injector devices A single 40-mg dose of Adalimumab was subcutaneously administered to healthy subjects.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — A single 40-mg dose of Adalimumab is administered subcutaneously to all the subjects.
  Other Names: CinnoRA; Humira

SUMMARY:
This study aims to demonstrate pharmacokinetic (PK) similarity of biosimilar candidate CinnoRA® relative to adalimumab reference product (Humira®) and evaluate safety and tolerability of CinnoRA®, in a parallel fashion in healthy volunteers after administration of a single dose (40 mg) of adalimumab.

The primary objective of this study is to demonstrate that the PK of CinnoRA® is similar to its originator, Humira®, as assessed by the area under the serum concentration time curve (AUC) from time 0 extrapolated to infinity (AUCinf) and the Cmax.

The secondary objectives of the study are:

* To further compare the PK of CinnoRA® and Humira®.
* To assess the safety of CinnoRA®.

DETAILED DESCRIPTION:
This is a single-dose trial with one administration of each product (CinnoRA® and Humira®). Each subject will participate in one treatment period, and will be randomised to receive CinnoRA® or Humira® in a parallel fashion. The subjects will be closely monitored during the following 24 hours (h), and will be allowed to leave the site in the next morning post evaluation and blood samples will be collected prior to and at the following time points after the dose: 4, 8, 12 and 24 hours post-dose (on day 2). The subjects will be requested to visit the trial site on days 3, 4, 5, 6, 7, 8, 9, 12, 15, 22, 29, 36, 43, 50, 57, 63 and 71 after dose for blood sampling and evaluation of safety variable and tolerability.

Before initiation, the trial is reviewed by food and drug administration of Iran. The protocol, case report form (CRF), information for subjects and informed consent form are submitted to the ethics committees responsible for review and approval purposes, according to national regulatory guidelines.

In this study, no subject is recruited without an informed consent. All the informed consent forms which are signed by the subjects have two copies so that subjects could receive a copy of it.

This is a single-dose trial with one administration of each product (CinnoRA® and Humira®). 74 (group A=37, group B=37) eligible subjects have been planned to enter to the study. All of whom are aged between 18 and 45 years. Subjects' randomization was done, using permuted block randomization method. Both groups received 40 mg of either of the drugs as a single subcutaneous injection. The injection method, injection pens and cartridges were totally the same in both groups. The primary objective of this study is to demonstrate that the PK of CinnoRA® is similar to its originator, Humira®, as assessed by the area under the serum concentration time curve (AUC) from time 0 extrapolated to infinity (AUCinf) and the Cmax. Secondary objectives include assessment of the time to Cmax (tmax), AUC from time 0 to the last quantifiable concentration (AUClast) of CinnoRA® compared with Humira®, as well as evaluation of safety and tolerability. The safety endpoints of the trial are to evaluate the incidence of reported adverse effects, detecting changes in vital signs, clinical laboratory tests (hematologic, biochemistry, urine analysis and urine culture tests) and ECG.

Determination of sample size:

An equivalence test of means AUCinf using two one-sided tests on data from a parallel-group design with sample sizes of 37 in the reference group and 37 in the treatment group achieves 81% power at a 10% significance level when the true ratio of the means AUCinf is 1.00, the coefficient of variation on the original, unlogged scale is 0.38, and the equivalence limits of the mean ratio AUCinf are 0.80 and 1.25.

DATA QUALITY ASSURANCE:

CinnaGen Company conducts clinical trials according to procedures that incorporate the ethical principles of GCP. Accurate and reliable data collection was assured by verification and cross-check of the CRFs against the subject's records by clinical monitors (source document verification was performed), and the maintenance of a drug-dispensing log by the center. A comprehensive validation check program was used to verify the data, and discrepancy reports were generated accordingly for resolution by the investigator.

Blinding:

This is a double-blind trial. During the clinical phase of the trial, neither the subjects nor the site personnel are aware of the identity (CinnoRA® and Humira®) of the treatments administered. However, there is an unblinded person who receives the randomisation list and dispenses the trial drugs according to the list. The unblinded person is not otherwise participate in the execution of the trial. The randomisation list determines the dispensing order of the trial products for each subject and only the randomisation number appear on the sample collection logs, as well as, on the sample aliquots delivered to the bioanalytical laboratory. Thus, the personnel responsible for analysing the PK samples are also be blinded.

Randomisation envelopes are stored in the ISF, in a locked cabinet. In a case of emergency, the code of an individual subject may be opened and the reasons for opening will be documented and the subject will be discontinued from the trial

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed ICF to participate in the trial and to comply with the trial procedures.
2. Be healthy male and female between the ages of 18 and 45 years. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, complete physical examination including blood pressure and heart rate measurement, 12 lead ECG and clinical laboratory tests.
3. Have a Body Mass Index (BMI) of 19.0 to 30.5 kg/m2;
4. Have Chest X ray with no evidence of current active TB or previous (inactive) TB, general infections, heart failure, malignancy, or other clinically significant abnormalities taken at Screening or within 24 weeks prior to Day 1 and read by a qualified radiologist.
5. Female subjects with child-bearing potential must agree to use a medically accepted method of contraception during the trial and one month after the end of the trial. Acceptable methods of contraception include the following:

   * Stable oral/transdermal/injectable hormonal contraceptive regimen without break through uterine bleeding and condom/spermicide.
   * Intrauterine device (inserted at least 2 months prior to screening visit) used with spermicide/condom.
   * Condom (male or female) with spermicide
   * Vasectomy of the male partner in conjunction with condom or spermicide.

Exclusion Criteria:

1. Being doubtful about their availability to complete the trial.
2. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic (Multiple sclerosis), autoimmune, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
3. Previous history of cancer, except for adequately treated basal cell or squamous cell carcinoma of the skin.
4. Active or latent Tuberculosis or who have a history of Tuberculosis
5. History of invasive systemic fungal infections or other opportunistic infections
6. Systemic or local infection, a known risk for developing sepsis and/or known active inflammatory process
7. Serious infection associated with hospitalisation and/or which required intravenous antibiotics
8. History of and/or current cardiac disease
9. Have received live vaccine(s) within 4 weeks prior to Screening or who will require live vaccine(s) between Screening and the final study visit
10. Intake medication with a half-life > 24 h within 4 weeks or 5 half-lives of the medication prior to investigational product administration
11. Have a history of smoking >10 cigarettes per day.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2016-10-22 (Actual); Primary Completion 2017-08-06 (Actual); Study Completion 2017-08-06 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to infinity (AUCinf) | 71 days
  AUCinf will be calculated using the equation:AUCinf= AUClast + (Clast / Kel)
Maximum serum concentration (Cmax) | 71 days
  It is obtained directly from the observed concentration-time data

SECONDARY OUTCOMES:
Area under the concentration-time curve from time zero to the last quantifiable concentration (AUClast) | 71 days
  It is calculated using the linear trapezoidal rule
Time to Cmax (Tmax) | 71 days
  It is obtained directly from the observed concentration-time data

CONTACTS AND LOCATIONS:
Overall Officials: Somayeh Amini, PharmD, Study Director — Orchid Pharmed Company
Locations (1):
- Orchidpharmed PK/PD site, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaur P, Chow V, Zhang N, Moxness M, Kaliyaperumal A, Markus R. A randomised, single-blind, single-dose, three-arm, parallel-group study in healthy subjects to demonstrate pharmacokinetic equivalence of ABP 501 and adalimumab. Ann Rheum Dis. 2017 Mar;76(3):526-533. doi: 10.1136/annrheumdis-2015-208914. Epub 2016 Jul 27. PMID 27466231
- [Background] Hyland E, Mant T, Vlachos P, Attkins N, Ullmann M, Roy S, Wagner V. Comparison of the pharmacokinetics, safety, and immunogenicity of MSB11022, a biosimilar of adalimumab, with Humira((R)) in healthy subjects. Br J Clin Pharmacol. 2016 Oct;82(4):983-93. doi: 10.1111/bcp.13039. Epub 2016 Jul 28. PMID 27285856
- [Background] Ma VY, Chan L, Carruthers KJ. Incidence, prevalence, costs, and impact on disability of common conditions requiring rehabilitation in the United States: stroke, spinal cord injury, traumatic brain injury, multiple sclerosis, osteoarthritis, rheumatoid arthritis, limb loss, and back pain. Arch Phys Med Rehabil. 2014 May;95(5):986-995.e1. doi: 10.1016/j.apmr.2013.10.032. Epub 2014 Jan 21. PMID 24462839
- [Background] Davatchi F, Jamshidi AR, Banihashemi AT, Gholami J, Forouzanfar MH, Akhlaghi M, Barghamdi M, Noorolahzadeh E, Khabazi AR, Salesi M, Salari AH, Karimifar M, Essalat-Manesh K, Hajialiloo M, Soroosh M, Farzad F, Moussavi HR, Samadi F, Ghaznavi K, Asgharifard H, Zangiabadi AH, Shahram F, Nadji A, Akbarian M, Gharibdoost F. WHO-ILAR COPCORD Study (Stage 1, Urban Study) in Iran. J Rheumatol. 2008 Jul;35(7):1384. Epub 2008 May 1. PMID 18464299
- [Background] Wong M, Ziring D, Korin Y, Desai S, Kim S, Lin J, Gjertson D, Braun J, Reed E, Singh RR. TNFalpha blockade in human diseases: mechanisms and future directions. Clin Immunol. 2008 Feb;126(2):121-36. doi: 10.1016/j.clim.2007.08.013. Epub 2007 Oct 3. PMID 17916444
- [Background] Wiens A, Correr CJ, Venson R, Otuki MF, Pontarolo R. A systematic review and meta-analysis of the efficacy and safety of adalimumab for treating rheumatoid arthritis. Rheumatol Int. 2010 Jun;30(8):1063-70. doi: 10.1007/s00296-009-1111-4. Epub 2009 Aug 26. PMID 19707765
- [Derived] Jamshidi A, Sabzvari A, Anjidani N, Shahpari R, Badri N. A randomized phase I pharmacokinetic trial comparing the potential biosimilar adalimumab (CinnoRA(R)) with the reference product (Humira(R)) in healthy volunteers. Expert Opin Investig Drugs. 2020 Mar;29(3):327-331. doi: 10.1080/13543784.2020.1723000. Epub 2020 Jan 30. PMID 31985294